CLINICAL TRIAL: NCT02078362
Title: Evaluation of Antibody-dependent Cell Cytotoxicity (ADCC) Against Gastric Cancer Cells
Brief Title: ADCC Against Gastric Cancer Cells
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Yong Wei Peng, National University Hospital, Singapore
Other Study IDs: KK002; 2013/00654 (Other: NHG Domain Specific Review Board)
Record Dates: First submitted 2013-12-09; First posted 2014-03-05 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Peripheral blood will be taken from the enrolled patients at National University Hospital and from healthy volunteers. ADCC assay will be performed for evaluating efficacy of new medicine candidates.

ELIGIBILITY:
Inclusion Criteria:

For the gastric cancer patients, patients with 21 years of age and above and younger than 80 years old who have gastric cancer can enroll in this study. For the healthy donors, healthy volunteers with 21 years of age and above and younger than 80 years old can enroll in this study.

Exclusion Criteria:

(A) Age of <21 and >80 years old (B) Pregnancy (C) Decision of unsuitableness by Principal Investigator or physician-in-charge

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastric cancer patients treated at National University Hospital.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of cell lysis | within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wei Peng Yong, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Macdonald JS, Smalley SR, Benedetti J, Hundahl SA, Estes NC, Stemmermann GN, Haller DG, Ajani JA, Gunderson LL, Jessup JM, Martenson JA. Chemoradiotherapy after surgery compared with surgery alone for adenocarcinoma of the stomach or gastroesophageal junction. N Engl J Med. 2001 Sep 6;345(10):725-30. doi: 10.1056/NEJMoa010187. PMID 11547741